CLINICAL TRIAL: NCT06205680
Title: Soft Mist Nasal Administration Device for Topical Anaesthesia of the Nasal Cavity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: CT1 NAA lido
Record Dates: First submitted 2023-12-27; First posted 2024-01-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Participants are not randomized. A randomization (paper) strategy will be applied to determine which drug will be applied in which nostril
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAA with Lidocaine (Experimental): One 1 ml syringes with lidocaine 2 % will be prepared and connected to the NAA device. The device will be placed in front of a nostril and the subject is asked not to breath until 0,5 ml of lidocaine has been administered. The lidocaine will be sprayed by the attending anaesthesiologist. After a waiting period of 2 minutes another 0,5 ml of lidocaine will be administered (= total of 1 ml lidocaine 2%).
  Interventions: Device: NAA for topical anaesthesia of the nasal cavity
- NAA with NaCl 0,9% (Experimental): One 1 ml syringes with NaCl 0,9 % will be prepared and connected to the NAA device.
  The device will be placed in front of the other nostril and the subject is asked not to breath until 0,5 ml of NaCl has been administered. The NaCl will be sprayed by the attending anaesthesiologist. After a waiting period of 2 minutes another 0,5 ml of NaCl will be administered (= total of 1 ml NaCl 0,9%).
  Interventions: Device: NAA for topical anaesthesia of the nasal cavity

INTERVENTIONS:
Device: NAA for topical anaesthesia of the nasal cavity — NAA for topical anaesthesia of the nasal cavity

SUMMARY:
Rationale:

Effective and fast topical anesthesia of the nasal mucosa is of paramount importance for nasal instrumentation like nasal fiberoptic procedures, awake nasal fiberoptic intubation and placement of nasogastric tubes. Conventional topical anesthesia for the nasal mucosa is often patchy and not always effective. The investigators hypothesize that topical anesthesia of the nasal mucosa with the nasal atomizer adapter (NAA) provides good to excellent nasal topical anesthesia with high patient comfort.

Objective: In this study the NAA will be used for nasal topical anesthesia. The investigators will evaluate complete anesthesia of the nasal mucosa for nasal instrumentation, the use of the NAA and the comfort level for the subjects.

Study design: Interventional study.

Study population: 20 healthy human volunteers, ASA 1, 18-60 years old.

Intervention: Lidocaine 2% will be applied intranasally with the NAA before nasal instrumentation. On completion of the procedure the participant and the researcher will be asked to complete a feedback form.

Main study parameters/endpoints:

Studying the level of anesthesia of the nasal mucosa as evaluated and demonstrated with successful awake nasal instrumentation with minimal discomfort for the subject.

Nature and extent of the burden and risks associated with participation:

Risk management on the nasal atomizer adapter (NAA) shows that all user risks are mitigated and no residual risks remain for the use of the device. Testing of the device and the application of the device in daily practice has no additional risks than the present technique of performing topical anaesthesia of the nasal mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years
* Lean body weight >= 50 kg
* ASA physical status 1

Exclusion Criteria:

* Inability to cooperate
* History of hepatic, renal and coagulation diseases,
* Respiratory tract pathology
* Obstruction of the nasal passage
* Chronic rhinitis
* Chronic sinusitis
* Pregnancy
* Allergy to amide type of local anaesthetics
* No written informed consent by subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Level of anesthesia | on day of intervention
  Studying the level of anesthesia of the nasal mucosa as evaluated and demonstrated with successful awake nasal instrumentation with minimal discomfort for the subject.

SECONDARY OUTCOMES:
Use of the NAA | on day of intervention
  The convenience of using the NAA, reported by using a questionnaire.
Comfort level of NAA | on day of intervention
  Studying the level of comfort of NAA for the patient, reported by using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Hielke Markerink, Study Director — Radboud University Medical Center (Radboudumc); Geerf-Jan van Geffen, Principal Investigator — Radboud University Medical Center (Radboudumc); Jörgen Bruhn, Study Chair — Radboud University Medical Center (Radboudumc)
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No